CLINICAL TRIAL: NCT02187705
Title: Observation of Therapy With Micardis® (Telmisartan) in Patients With Essential Hypertension in Hospitals
Brief Title: Micardis® in Patients With Essential Hypertension
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.322
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Patients with normotension at baseline
  Interventions: Drug: Telmisartan tablets
- Patients with essential hypertension at baseline
  Interventions: Drug: Telmisartan tablets
- Patients with isolated hypertension at baseline
  Interventions: Drug: Telmisartan tablets

INTERVENTIONS:
Drug: Telmisartan tablets — All patients were treated with different doses of telmisartan for 14 days
  Other Names: Micardis®

SUMMARY:
The aim of this observational study was to supplement the data on efficacy, safety, and tolerability of telmisartan under daily conditions in hospitals

ELIGIBILITY:
Inclusion Criteria:

* Patients with essential hypertension
* Minimum age of 18 years

Exclusion Criteria: Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1688 (Actual)
Dates: Start 1999-05; Primary Completion 2000-05 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in blood pressure | Up to 14 days
  Evaluation was performed separately for three patient groups depending on their hypertension status at baseline (normotension, essential hypertension and isolated hypertension)
Number of patients with adverse events | Up to 14 days